CLINICAL TRIAL: NCT05460026
Title: Effects Of Power Ball Exercises In Addition To Routine Physical Therapy On Pain, Grip Strength And Functional Disability In Patients With Carpal Tunnel Syndrome
Brief Title: Effects Of Power Ball Exercises In Addition To Routine Physical Therapy In Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muhammad Jahanzaib Rasool
Record Dates: First submitted 2022-07-01; First posted 2022-07-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Physical therapy; Median Neuropathy; Power Ball Exercise; Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be single blinded in which the assessor will be unaware of the treatment intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Routine physical therapy will be given to the participants of group A
  Interventions: Other: Routine Physical Therapy
- Group B (Experimental): Powerball exercises with routine physical therapy will be given to the participants of group B
  Interventions: Other: Powerball Exercises

INTERVENTIONS:
Other: Routine Physical Therapy — Participants will receive routine physical therapy which includes ultrasound, nerve gliding, tendon mobilization, stretching, mobility and strengthening exercises for the wrist. Each session will last for 30 minutes with 12 sessions on alternate days (3 sessions / week).
  Arms: Group A
Other: Powerball Exercises — Participants will be using the Powerball™ for 5 minutes per hand, 3 times a week along with routine physical therapy exercises.
  Arms: Group B

SUMMARY:
The purpose for doing this study is to determine that whether use of Power Ball in form of resistance training will be effective in increasing grip strength in carpel tunnel syndrome patient and possible benefits of the regime as effective means of rehabilitation for wrist and hand injuries. Moreover for increasing grip strength it can be used as an adjunct for physical therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 45-60 years
2. Both male and female
3. Clinically diagnosed carpal tunnel syndrome
4. Carpal Tunnel Syndrome for a duration of more than 02 months
5. Tingling sensation and numbness over the dorsal surface of thumb, index, middle, and lateral 1/3rd of ring fingers
6. Positive Tinel's sign
7. Positive Phalen's Maneuver

Exclusion Criteria:

1. Any previous trauma, fracture, subluxation, dislocation, surgery or bony abnormalities around wrist joint in the past 5 years.
2. Symptomatic Arthritis of wrist joint
3. Cervical radiculopathy
4. Corticosteroid injection within 3 months

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change in pain will be measured at initial visit, at sixth session and at the twelfth session.
  Pain Intensity will be measured by Numeric Rating Scale (NRS)
Grip Strength | Change in grip strength will be measured at initial visit, at sixth session and at the twelfth session.
  Grip Strength will be measured by using handheld dynamometry (HHD)
Functional Disability | Change in functional disability will be measured at initial visit, at sixth session and at the twelfth session.
  Functional disability will be measured by Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Ahmed, PhD, Study Director — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Immediately after publication
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending on 36th month